CLINICAL TRIAL: NCT02590640
Title: Insular Inhibitory Neuromodulation to Reduce Cigarette Craving and Alter Brain Function in Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15-1016
Record Dates: First submitted 2015-10-26; First posted 2015-10-29 (Estimated); Results first posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-06

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhibitory insular rTMS (Active Comparator): Inhibitory (1 Hz) repetitive transcranial magnetic stimulation will be applied to the insula in smokers.
  Interventions: Device: Repetitive transcranial magnetic stimulation, MagStim Rapid2
- Sham insular rTMS (Sham Comparator): Sham repetitive transcranial magnetic stimulation will be applied to the insula in smokers.
  Interventions: Device: Sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation, MagStim Rapid2 — This study plans to learn more about the way an experimental technique called "transcranial magnetic stimulation" (TMS) affects a specific part of the brain, called the insula. Some research suggests that this part of the brain plays an important role in craving. The investigators plan to study the effects of TMS using standard surveys and magnetic resonance imaging (MRI) of subjects' brain.
  Arms: Inhibitory insular rTMS
Device: Sham repetitive transcranial magnetic stimulation — Sham repetitive transcranial magnetic stimulation will be applied to the insula in smokers.
  Arms: Sham insular rTMS

SUMMARY:
The goal of this study is to determine if a specific experimental brain stimulation technique can be used as a non-invasive way to reduce cigarette cravings in current smokers. This study plans to learn more about the way an experimental technique called "transcranial magnetic stimulation" (TMS) affects a specific part of the brain, called the insula. Some research suggests that this part of the brain plays an important role in craving. The investigators plan to study the effects of TMS using standard surveys and magnetic resonance imaging (MRI) of subjects' brain.

For interested participants, this study requires a single 3 hour appointment, which will include MRI of the brain as well as TMS.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55
2. Ability to provide informed consent
3. Self-reported current average daily cigarette consumption >10/day for at least 1 year
4. Self-reported motivation to quit smoking

Exclusion Criteria:

1. MRI/TMS exclusions, including

   * Claustrophobia
   * Intracranial or spinal hardware
   * Pacemakers
   * MR-incompatible devices (Examples: pacemaker, deep brain stimulator, vagal nerve stimulator, cochlear implant, insulin pump, implanted medication pump, bone stimulator, implanted defibrillator)
   * History of metal objects or fragments in the eye or skull, including shrapnel or metal plates
   * History of stroke or other brain lesion
   * History of attempted suicide or suicidal ideation
   * Personal history of headaches, seizures, epilepsy, or status epilepticus
   * Family history of epilepsy
   * Medications known to lower seizure threshold (e.g., tricyclic antidepressants, antipsychotics, psychostimulants)
   * Increased intracranial pressure, hydrocephalus, or pseudotumor cerebri
   * Unstable coronary artery disease
   * Current pregnancy or positive urine pregnancy test
2. Neurological illness
3. Prior neurosurgery
4. Schizophrenia
5. Bipolar disorder
6. Current (within the last two months) major depressive disorder
7. Substance dependence or positive urinalysis for opiates, stimulants, cannabis, or sedative on the day of testing
8. Alcohol dependence or positive breath test for alcohol on the day of testing
9. Use of tobacco products other than cigarettes.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11; Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Regner, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Department of Radiology, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Arms cannot be reported separately. Data for this study was found to have been compromised. The PI responsible for the study has left the institution, and the data regarding randomization, outcome measures, and adverse events has been determined to be unreliable.
Groups:
- All Participants: Inhibitory insular rTMS group: Inhibitory (1 Hz) repetitive transcranial magnetic stimulation will be applied to the insula in smokers. Repetitive transcranial magnetic stimulation, MagStim Rapid2:
  And
  Sham insular rTMS group: Sham repetitive transcranial magnetic stimulation will be applied to the insula in smokers.
Period: Overall Study
Arm/Group | All Participants
Started | 40
Completed | 37
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Arms cannot be reported separately. Data for this study was found to have been compromised. The PI responsible for the study has left the institution, and the data regarding randomization, outcome measures, and adverse events has been determined to be unreliable.
Arm/Group | All Participants
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 30
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Changes in Cue-induced Cigarette Craving (Post-treatment - Pre-treatment) as Assessed by TCQ
Description: Cue-induced cigarette craving as assessed by Tobacco Craving Questionnaire (TCQ)
Time Frame: 1 hour
Population: Data cannot be reported. Data for this study was found to have been compromised. The PI responsible for the study has left the institution, and the data regarding randomization, outcome measures, and adverse events has been determined to be unreliable.
Arm/Group | Inhibitory Insular rTMS | Sham Insular rTMS
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Changes in Craving Cue-induced fMRI Activity (Post-treatment - Pre-treatment) at Whole Brain Level Using Statistical Parametric Mapping
Time Frame: 1 hour
Population: as for outcome 1
Arm/Group | Inhibitory Insular rTMS | Sham Insular rTMS
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Changes in fMRI Connectivity (Post-treatment - Pre-treatment) at Whole Brain Level Using Statistical Parametric Mapping
Time Frame: 1 hour
Population: as for outcome 1
Arm/Group | Inhibitory Insular rTMS | Sham Insular rTMS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 day
Description: Arms cannot be reported separately, nor can data be reported. Data for this study was found to have been compromised. The PI responsible for the study has left the institution, and the data regarding randomization, outcome measures, and adverse events has been determined to be unreliable.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Data for this study was found to have been compromised. The P.I. responsible for the study has left the institution, and the data regarding randomization, outcome measures, and adverse events has been determined to be unreliable and cannot be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT02590640/Prot_SAP_000.pdf